CLINICAL TRIAL: NCT00995150
Title: A Phase 3, Multi-Center, Open-Label Study of a Levonorgestrel-Releasing Intrauterine System for Long-Term, Reversible Contraception
Brief Title: A Study of a Levonorgestrel-Releasing Intrauterine System for Long-Term, Reversible Contraception
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The data cutoff date of 05 April 2021 was chosen as it coincides with all subjects completing through Year 8 of use (intended duration of use for the product).
Sponsor: Medicines360 (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: M360-L102
Record Dates: First submitted 2009-10-13; First posted 2009-10-15 (Estimated); Results first posted 2024-08-14 (Actual); Last update posted 2024-08-14 (Actual); Status verified 2024-07

CONDITIONS: Contraception
Keywords: contraception; intrauterine; long-term; reversible
MeSH Terms: interventions — Levonorgestrel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- LNG20 (16-35 Year Olds) (Experimental): LNG20 levonorgestrel-releasing intrauterine system in subjects 16-35 years of age
  Interventions: Drug: LNG20
- Mirena (Active Comparator): Levonorgestrel-releasing intrauterine system for contraception
  Interventions: Drug: Mirena
- LNG20 (36-45 Year Olds) (Experimental): LNG20 levonorgestrel-releasing intrauterine system in subjects 36-45 years of age
  Interventions: Drug: LNG20

INTERVENTIONS:
Drug: LNG20 — levonorgestrel-releasing intrauterine system for contraception
  Other Names: Liletta
  Arms: LNG20 (16-35 Year Olds); LNG20 (36-45 Year Olds)
Drug: Mirena — Mirena intrauterine system
  Arms: Mirena

SUMMARY:
The primary objective of this study is to assess the efficacy of a levonorgestrel-releasing intrauterine system (LNG20) in nulliparous and parous females of child-bearing potential who request long-term, reversible contraception for up to 10 years.

DETAILED DESCRIPTION:
This is a Phase 3, randomized, open-label, multicenter evaluation of the efficacy of a levonorgestrel-releasing intrauterine system (LNG20). The goals of the study include provision of information to understand efficacy and safety within the widest range of possible users of the LNG20. Typically, intrauterine contraceptive studies only include women 18-35 years of age for efficacy and safety, and place limits on parity and larger body size. Women outside of these characteristics also desire an effective intrauterine contraceptive. Accordingly, this study will include women who are both nulliparous and parous as well as women less than 18 years of age in the primary efficacy and safety analyses

ELIGIBILITY:
Inclusion Criteria:

* Healthy women requesting contraception
* 16-35 years old
* Cohort 36-45 years old
* Sexually active

Exclusion Criteria:

* Currently pregnant, pregnant within 4 weeks prior to study entry or planning pregnancy within 24 months of study entry
* Currently breastfeeding
* Current persistent, abnormal vaginal bleeding

Ages: 16 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 1910 (Actual)
Dates: Start 2009-11 (Actual); Primary Completion 2021-10-12 (Actual); Study Completion 2021-10-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Olariu, MD, PhD, Study Director — COO
Locations (25):
- United States (25):
  - Phoenix, Arizona
  - Palo Alto, California
  - San Francisco, California
  - Vista, California
  - Denver, Colorado
  - Atlanta, Georgia
  - Idaho Falls, Idaho
  - Chicago, Illinois
  - Des Moines, Iowa
  - Ann Arbor, Michigan
  - St Louis, Missouri
  - New York, New York
  - Chapel Hill, North Carolina
  - Cincinnati, Ohio
  - Cleveland, Ohio
  - Columbus, Ohio
  - Tulsa, Oklahoma
  - Portland, Oregon
  - Philadelphia, Pennsylvania
  - Magee Women's Hospital, University of Pittsburgh, Pittsburgh, Pennsylvania
  - Dallas, Texas
  - Houston, Texas
  - Salt Lake City, Utah
  - Norfolk, Virginia
  - Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chen BA, Kimble T, Harris LH, Kerns JL, Olariu AI, Creinin MD. Levonorgestrel 52-mg Intrauterine Device Efficacy and Safety After More Than 8 Years of Use. Obstet Gynecol. 2023 May 1;141(5):1004-1006. doi: 10.1097/AOG.0000000000005147. Epub 2023 Apr 5. PMID 37023451
- [Derived] Chen BA, Eisenberg DL, Schreiber CA, Turok DK, Olariu AI, Creinin MD. Bleeding changes after levonorgestrel 52-mg intrauterine system insertion for contraception in women with self-reported heavy menstrual bleeding. Am J Obstet Gynecol. 2020 Apr;222(4S):S888.e1-S888.e6. doi: 10.1016/j.ajog.2019.11.1288. Epub 2019 Dec 19. PMID 31866516
- [Derived] Teal SB, Turok DK, Chen BA, Kimble T, Olariu AI, Creinin MD. Five-Year Contraceptive Efficacy and Safety of a Levonorgestrel 52-mg Intrauterine System. Obstet Gynecol. 2019 Jan;133(1):63-70. doi: 10.1097/AOG.0000000000003034. PMID 30531565
- [Derived] Schreiber CA, Teal SB, Blumenthal PD, Keder LM, Olariu AI, Creinin MD. Bleeding patterns for the Liletta(R) levonorgestrel 52 mg intrauterine system. Eur J Contracept Reprod Health Care. 2018 Apr;23(2):116-120. doi: 10.1080/13625187.2018.1449825. Epub 2018 Mar 21. PMID 29560743
- [Derived] Darney PD, Stuart GS, Thomas MA, Cwiak C, Olariu A, Creinin MD. Amenorrhea rates and predictors during 1 year of levonorgestrel 52 mg intrauterine system use. Contraception. 2018 Mar;97(3):210-214. doi: 10.1016/j.contraception.2017.10.005. Epub 2017 Oct 13. PMID 29038072
- [Derived] Creinin MD, Jansen R, Starr RM, Gobburu J, Gopalakrishnan M, Olariu A. Levonorgestrel release rates over 5 years with the Liletta(R) 52-mg intrauterine system. Contraception. 2016 Oct;94(4):353-6. doi: 10.1016/j.contraception.2016.04.010. Epub 2016 Apr 25. PMID 27125892
- [Derived] Eisenberg DL, Schreiber CA, Turok DK, Teal SB, Westhoff CL, Creinin MD; ACCESS IUS Investigators. Three-year efficacy and safety of a new 52-mg levonorgestrel-releasing intrauterine system. Contraception. 2015 Jul;92(1):10-6. doi: 10.1016/j.contraception.2015.04.006. Epub 2015 Apr 28. PMID 25934164

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Enrollment into the Mirena arm was stopped when it was determined that sufficient comparative safety data for LILETTA vs. Mirena was already available; thereafter, subjects were only assigned to LILETTA. The data cutoff date of 05 April 2021 was chosen for all LILETTA subjects as it coincides with all subjects completing through Year 8 of use (intended duration of use for the product). All Mirena participants were discontinued by the end of Year 5.
Groups:
- LNG20 (16-35 Yr Olds): LNG20 levonorgestrel-releasing intrauterine system
  LNG20: levonorgestrel-releasing intrauterine system for contraception sub-population (16-35 years old)
- LNG20 (36-45 Yr Olds): LNG20 levonorgestrel-releasing intrauterine system
  LNG20: levonorgestrel-releasing intrauterine system for contraception sub-population (36-45 years old)
Period: Overall Study
Arm/Group | LNG20 (16-35 Yr Olds) | Mirena | LNG20 (36-45 Yr Olds)
Started | 1600 | 159 | 151
Completed | 302 | 22 | 41
Not Completed | 1298 | 137 | 110

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | LNG20 (16-35 Yr Olds) | Mirena | LNG20 (36-45 Yr Olds) | Total
Number analyzed (Participants) | 1600 | 159 | 151 | 1910
Age, Customized [Count of Participants; unit: Participants]
  Age 16-35 years | 1,600 | 159 | 0 | 1759
  Age 36-45 years | 0 | 0 | 151 | 151
Age, Customized [Mean (Standard Deviation); unit: years] | 26.2 (4.4) | 26.1 (4.4) | 39.6 (2.7) | 27.2 (5.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1600 | 159 | 151 | 1910
  Male | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 237 | 21 | 21 | 279
  Not Hispanic or Latino | 1363 | 138 | 130 | 1631
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 19 | 2 | 2 | 23
  Asian | 61 | 5 | 7 | 73
  Native Hawaiian or Other Pacific Islander | 5 | 0 | 1 | 6
  Black or African American | 212 | 12 | 20 | 244
  White | 1250 | 131 | 120 | 1501
  More than one race | 49 | 8 | 1 | 58
  Unknown or Not Reported | 4 | 1 | 0 | 5
BMI [Count of Participants; unit: Participants]
  BMI ≤24.9 | 823 | 68 | 59 | 950
  BMI 25-29.9 | 390 | 52 | 37 | 479
  BMI 30-39.9 | 304 | 28 | 41 | 373
  BMI ≥40 | 79 | 11 | 14 | 104
  No Weight Taken at Baseline | 4 | 0 | 0 | 4
Partner Status [Count of Participants; unit: Participants]
  Lives with Partner | 915 | 84 | 106 | 1105
  Does Not Live with Partner | 685 | 75 | 45 | 805
Parity [Count of Participants; unit: Participants]
  Nulliparous | 989 | 90 | 22 | 1101
  Parous | 611 | 69 | 129 | 809
BMI [Mean (Standard Deviation); unit: (kg/m^2)] — Population: 4 participants' weights in the LNG20 (16-35 year olds) arm were not measured at baseline and therefore were not analyzed in the mean
  (kg/m^2)
    number analyzed (Participants) | 1596 | 159 | 151 | 1906
    (all) | 26.8 (6.7) | 27.2 (6.7) | 28.6 (7.6) | 26.9 (6.8)

OUTCOME MEASURES:

1. Primary Outcome: Number of Pregnancies Per Year
Description: Number of pregnancies per year in each treatment arm.
Time Frame: 10 years
Population: All Mirena participants were discontinued by end of Year 5; therefore, Years 6-10 are considered "not available" for that arm.
Measure: Number; unit: pregnancies
Groups:
- LNG20 (16-35 Yr Olds): LNG20 levonorgestrel-releasing intrauterine system
  LNG20: levonorgestrel-releasing intrauterine system for contraception (16-35 Yr Olds)
- Mirena: Levonorgestrel-releasing intrauterine system for contraception Mirena: Mirena intrauterine system
Arm/Group | LNG20 (16-35 Yr Olds) | Mirena | LNG20 (36-45 Yr Olds)
Number analyzed (Participants) | 1600 | 159 | 151
pregnancies
  Year 1 | 2 | 1 | 0
  Year 2 | 4 | 0 | 0
  Year 3 | 1 | 0 | 0
  Year 4 | 1 | 0 | 0
  Year 5 | 1 | 1 | 0
  Year 6 | 0 | NA — All Mirena participants were discontinued by end of Year 5. | 0
  Year 7 | 2 | NA — All Mirena participants were discontinued by end of Year 5. | 0
  Year 8 | 0 | NA — All Mirena participants were discontinued by end of Year 5. | 0
  Year 9 | 0 | NA — All Mirena participants were discontinued by end of Year 5. | 0
  Year 10 | 0 | NA — All Mirena participants were discontinued by end of Year 5. | 0

2. Primary Outcome: Cumulative Pearl Index
Description: The Pearl Index (PI) is an estimate of the number of pregnancies per 100 women-years of contraceptive exposure. The Pearl Index is calculated as the number of "on treatment" pregnancies in the study divided by the total number of complete 28-day cycles of use in the study multiplied by 1,300 (13 cycles/yr x 100 years). Cycles where other birth control methods were used were excluded from this measure. The Pearl Index for MIRENA was not a pre-specified primary outcome measure and is therefore not included. There is only 8 years of data due to the early termination of the study.
Time Frame: 8 years
Population: The Pearl Index for MIRENA was not a pre-specified primary outcome measure and is therefore not included. The number of participants analyzed for this measure is the MITT population.
Measure: Number (95% Confidence Interval); unit: pregnancies per 100 women-years
Arm/Group | LNG20 (16-35 Yr Olds) | LNG20 (36-45 Yr Olds)
Number analyzed (Participants) | 1538 | 146
pregnancies per 100 women-years
  Year 1 | 0.15 [0.02 to 0.55] | 0.0 [0 to 2.83]
  Year 2 | 0.25 [0.09 to 0.54] | 0.0 [0 to 1.49]
  Year 3 | 0.21 [0.08 to 0.43] | 0.0 [0 to 1.04]
  Year 4 | 0.20 [0.08 to 0.39] | 0.0 [0 to 0.81]
  Year 5 | 0.19 [0.09 to 0.36] | 0.0 [0 to 0.67]
  Year 6 | 0.17 [0.08 to 0.33] | 0.0 [0 to 0.59]
  Year 7 | 0.19 [0.10 to 0.35] | 0.0 [0 to 0.52]
  Year 8 | 0.19 [0.09 to 0.33] | 0.0 [0 to 0.48]

3. Secondary Outcome: Safety and Tolerability
Description: The safety and tolerability based on the report of adverse events and serious adverse events
Time Frame: 10 Years
Population: All Mirena participants were discontinued by end of Year 5.
Measure: Count of Participants; unit: Participants
Arm/Group | LNG20 (16-35 Yr Olds) | Mirena | LNG20 (36-45 Yr Olds)
Number analyzed (Participants) | 1600 | 159 | 151
Participants
  Subjects Reporting at Least One AE | 1441 | 138 | 137
  Subjects Reporting at Least One SAE | 79 | 6 | 8
  Subjects Reporting No AE or SAE | 80 | 15 | 6

4. Secondary Outcome: Distribution of Bleeding Amenorrhea by 90 Day Interval
Description: The incidence of diary reported bleeding and/or spotting by 90-day interval, as an assessment of IUS-induced amenorrhea, is summarized as the number of subjects reporting no bleeding and/or spotting.
Time Frame: 8 Years
Population: All Mirena participants were discontinued by end of Year 5.
Measure: Count of Participants; unit: Participants
Arm/Group | LNG20 (16-35 Yr Olds) | Mirena | LNG20 (36-45 Yr Olds)
Number analyzed (Participants) | 1600 | 159 | 151
Participants
  90 Day Interval 1 (Month 3): number analyzed (Participants) | 1554 | 153 | 146
  90 Day Interval 1 (Month 3) | 6 | 0 | 1
  90 Day Interval 2 (Month 6): number analyzed (Participants) | 1478 | 140 | 143
  90 Day Interval 2 (Month 6) | 167 | 27 | 16
  90 Day Interval 4 (Month 12): number analyzed (Participants) | 1320 | 123 | 128
  90 Day Interval 4 (Month 12) | 250 | 26 | 19
  90 Day Interval 8 (Month 24): number analyzed (Participants) | 1062 | 81 | 114
  90 Day Interval 8 (Month 24) | 283 | 27 | 35
  90 Day Interval 12 (Month 36): number analyzed (Participants) | 876 | 65 | 105
  90 Day Interval 12 (Month 36) | 319 | 21 | 40
  90 Day Interval 16 (Month 48): number analyzed (Participants) | 743 | 51 | 97
  90 Day Interval 16 (Month 48) | 275 | 23 | 37
  90 Day Interval 20 (Month 60): number analyzed (Participants) | 618 | 38 | 89
  90 Day Interval 20 (Month 60) | 249 | 16 | 35
  90 Day Interval 24 (Month 72): number analyzed (Participants) | 509 | 0 | 78
  90 Day Interval 24 (Month 72) | 199 |  | 33
  90 Day Interval 28 (Month 84): number analyzed (Participants) | 417 | 0 | 72
  90 Day Interval 28 (Month 84) | 157 |  | 33
  90 Day Interval 32 (Month 96): number analyzed (Participants) | 304 | 0 | 61
  90 Day Interval 32 (Month 96) | 115 |  | 28

5. Secondary Outcome: Continuation Rates
Description: The rate of continuation of usage over time.
Time Frame: 10 Years
Population: All Mirena participants were discontinued by the end of Year 5 per the study protocol. All LNG20 (36-45 Yr Old) participants were discontinued by the end of Year 8 per the study protocol. Month 6 is defined as 182 days of use, Year 1= 365 days, Year 2= 730 days, Year 3= 1095 days, Year 4= 1460 days, Year 5= 1825 days, Year 6= 2190 days, Year 7= 2555 days, Year 8= 2920 days, Year 9= 3285 days, and Year 10= 3650 days of product use.
Measure: Count of Participants; unit: Participants
Arm/Group | LNG20 (16-35 Yr Olds) | Mirena | LNG20 (36-45 Yr Olds)
Number analyzed (Participants) | 1600 | 159 | 151
Participants
  Number of Subjects Continuing Through Month 6 | 1420 | 131 | 133
  Number of Subjects Continuing Month 6 Through Year 1 | 1275 | 118 | 125
  Number of Subjects Continuing Year 1 Through Year 2 | 1034 | 86 | 114
  Number of Subjects Continuing Year 2 Through Year 3 | 859 | 64 | 105
  Number of Subjects Continuing Year 3 Through Year 4 | 720 | 49 | 98
  Number of Subjects Continuing Year 4 Through Year 5 | 597 | 21 | 91
  Number of Subjects Continuing Year 5 Through Year 6: number analyzed (Participants) | 1600 | 0 | 151
  Number of Subjects Continuing Year 5 Through Year 6 | 498 | 0 | 77
  Number of Subjects Continuing Year 6 Through Year 7: number analyzed (Participants) | 1600 | 0 | 151
  Number of Subjects Continuing Year 6 Through Year 7 | 402 | 0 | 72
  Number of Subjects Continuing Year 7 Through Year 8: number analyzed (Participants) | 1600 | 0 | 151
  Number of Subjects Continuing Year 7 Through Year 8 | 293 | 0 | 39
  Number of Subjects Continuing Year 8 Through Year 9: number analyzed (Participants) | 1600 | 0 | 151
  Number of Subjects Continuing Year 8 Through Year 9 | 83 | 0 | 0
  Number of Subjects Continuing Year 9 Through Year 10: number analyzed (Participants) | 1600 | 0 | 0
  Number of Subjects Continuing Year 9 Through Year 10 | 76 | 0 | 0

6. Secondary Outcome: Return of Menses After Discontinuation
Description: Subjects who discontinued from the trial and who were not pregnant or did not start a hormonal contraceptive were followed to assess the return of menses after IUS removal. If after three months menses had not occurred, the subject was to be evaluated for the cause of their secondary amenorrhea and continued to be followed monthly until the diagnosis was established.
Time Frame: 5 months
Population: Only those subjects who completed this evaluation are included.
Measure: Count of Participants; unit: Participants
Arm/Group | LNG20 (16-35 Yr Olds) | Mirena | LNG20 (36-45 Yr Olds)
Number analyzed (Participants) | 664 | 49 | 48
Participants
  Number (%) of Subjects With Onset of Menses Post-IUS Removal | 651 | 46 | 38
  Month 1 | 492 | 37 | 22
  Month 2 | 141 | 8 | 15
  Month 3 | 15 | 1 | 0
  Month 4 | 1 | 0 | 1
  Month 5 | 2 | 0 | 0

7. Secondary Outcome: Return to Fertility After Discontinuation
Description: Subjects who discontinued from the trial and desired pregnancy were followed for up to 12 months to assess fertility after IUS removal.
Time Frame: 12 months
Population: Distribution of Pregnancies (Months Post-IUS Removal) [N(%)]
Measure: Count of Participants; unit: Participants
Groups:
- Mirena: LNG20: levonorgestrel-releasing intrauterine system for contraception sub-population (16-35 years old) Levonorgestrel-releasing intrauterine system for contraception Mirena: Mirena intrauterine system
Arm/Group | LNG20 (16-35 Yr Olds) | Mirena | LNG20 (36-45 Yr Olds)
Number analyzed (Participants) | 241 | 19 | 3
Participants
  Total Number of Participants Pregnant | 201 | 15 | 2
  Month 1: number analyzed (Participants) | 201 | 15 | 2
  Month 1 | 17 | 3 | 0
  Month 2: number analyzed (Participants) | 201 | 15 | 2
  Month 2 | 36 | 5 | 0
  Month 3: number analyzed (Participants) | 201 | 15 | 2
  Month 3 | 34 | 2 | 0
  Month 4: number analyzed (Participants) | 201 | 15 | 2
  Month 4 | 28 | 0 | 0
  Month 5: number analyzed (Participants) | 201 | 15 | 2
  Month 5 | 20 | 2 | 1
  Month 6: number analyzed (Participants) | 201 | 15 | 2
  Month 6 | 18 | 1 | 0
  Month 7: number analyzed (Participants) | 201 | 15 | 2
  Month 7 | 15 | 0 | 0
  Month 8: number analyzed (Participants) | 201 | 15 | 2
  Month 8 | 16 | 1 | 0
  Month 9: number analyzed (Participants) | 201 | 15 | 2
  Month 9 | 6 | 0 | 0
  Month 10: number analyzed (Participants) | 201 | 15 | 2
  Month 10 | 5 | 1 | 1
  Month 11: number analyzed (Participants) | 201 | 15 | 2
  Month 11 | 5 | 0 | 0
  Month 12: number analyzed (Participants) | 201 | 15 | 2
  Month 12 | 1 | 0 | 0

8. Secondary Outcome: Mean Plasma Levonorgestrel Concentrations (pg/mL) for Subjects in the PK Substudy
Description: The Mean Plasma Pharmacokinetics of LNG in a Subset of Subjects through 60 Months of Use. "Non-obese" was defined as a BMI less than 30 kg/m^2. "Obese" was defined as a BMI of 30 kg/m^2 or higher.
Time Frame: 5 Years
Population: Mean Plasma Levonorgestrel Concentrations (pg/mL) for All Subjects in the PK Substudy.
Measure: Mean (Standard Deviation); unit: (pg/mL)
Groups:
- LNG20 (Obese): LNG20 levonorgestrel-releasing intrauterine system LNG20: levonorgestrel-releasing intrauterine system for contraception sub-population (obese)
- Mirena (Non-Obese): Levonorgestrel-releasing intrauterine system for contraception
  Mirena: Mirena intrauterine system (Non-Obese)
- LNG20 (Non-Obese): LNG20 levonorgestrel-releasing intrauterine system LNG20: levonorgestrel-releasing intrauterine system for contraception sub-population (Non-Obese)
Arm/Group | LNG20 (Obese) | Mirena (Non-Obese) | LNG20 (Non-Obese)
Number analyzed (Participants) | 19 | 18 | 21
(pg/mL)
  Week 1 | 187.6 (53.4) | 328.9 (150) | 310 (139.7)
  Week 2 | 199.3 (59) | 320.3 (147.4) | 278.7 (107)
  Month 1: number analyzed (Participants) | 19 | 17 | 21
  Month 1 | 180.5 (44.8) | 251 (98.2) | 247.7 (82.6)
  Month 3: number analyzed (Participants) | 17 | 17 | 21
  Month 3 | 166.8 (40.8) | 222.7 (58.5) | 237.4 (75)
  Month 6: number analyzed (Participants) | 17 | 16 | 20
  Month 6 | 153.7 (40) | 215.8 (59) | 229.5 (67.3)
  Month 9: number analyzed (Participants) | 15 | 14 | 19
  Month 9 | 134.9 (38.4) | 184.9 (52.4) | 229.9 (69.9)
  Month 12: number analyzed (Participants) | 16 | 13 | 18
  Month 12 | 140.5 (52.6) | 182.5 (43.9) | 192.3 (36.2)
  Month 18: number analyzed (Participants) | 14 | 11 | 16
  Month 18 | 126.3 (32.6) | 168.1 (32.1) | 168.6 (38.5)
  Month 24: number analyzed (Participants) | 15 | 9 | 17
  Month 24 | 115.7 (26.6) | 150.2 (28.9) | 180.8 (39.9)
  Month 30: number analyzed (Participants) | 14 | 8 | 13
  Month 30 | 111.1 (33.2) | 161.1 (51.3) | 164.2 (43.5)
  Month 36: number analyzed (Participants) | 12 | 6 | 11
  Month 36 | 104 (53.9) | 152.3 (50.5) | 152.6 (38.4)
  Month 42: number analyzed (Participants) | 9 | 6 | 13
  Month 42 | 101.7 (43.9) | 131 (51) | 151.9 (41.8)
  Month 48: number analyzed (Participants) | 8 | 5 | 11
  Month 48 | 93.2 (30.6) | 114.5 (33.8) | 136.1 (37.9)
  Month 54: number analyzed (Participants) | 5 | 2 | 11
  Month 54 | 93.7 (22.3) | 103.3 (43.5) | 127.3 (40.8)
  Month 60: number analyzed (Participants) | 6 | 2 | 10
  Month 60 | 68.1 (30.3) | 136.9 (62.4) | 109.5 (34.9)

9. Secondary Outcome: Plasma LNG Levels in All Subjects With Continuing Use From Month 36 Through Month 120
Description: The Plasma LNG Levels in All Subjects With Continuing Use From Month 36 Through Month 120.
Time Frame: month 36 through 120
Population: Plasma Levonorgestrel Concentrations for All Subjects Beginning at Month 36. All Mirena participants were discontinued by the end of Year 5.
Measure: Mean (Standard Deviation); unit: Levonorgestrel Concentration (pg/mL)
Arm/Group | LNG20 (16-35 Yr Olds) | Mirena | LNG20 (36-45 Yr Olds)
Number analyzed (Participants) | 810 | 62 | 104
Levonorgestrel Concentration (pg/mL)
  Month 36 | 129.879 (49.793) | 141.175 (60.438) | 152.693 (76.452)
  Month 42: number analyzed (Participants) | 740 | 55 | 98
  Month 42 | 117.907 (46.533) | 142.036 (73.278) | 155.518 (96.174)
  Month 48: number analyzed (Participants) | 703 | 50 | 90
  Month 48 | 110.109 (47.046) | 136.894 (97.898) | 141.066 (73.341)
  Month 54: number analyzed (Participants) | 607 | 39 | 91
  Month 54 | 105.095 (43.37) | 113.836 (40.715) | 140.576 (81.446)
  Month 60: number analyzed (Participants) | 520 | 37 | 88
  Month 60 | 97.721 (38.819) | 111.676 (49.42) | 118.826 (55.593)
  Month 66: number analyzed (Participants) | 300 | 0 | 72
  Month 66 | 94.284 (34.73) |  | 102.41 (43.507)
  Month 72: number analyzed (Participants) | 193 | 0 | 50
  Month 72 | 89.805 (42.318) |  | 98.542 (47.527)
  Month 78: number analyzed (Participants) | 151 | 0 | 45
  Month 78 | 87.897 (32.714) |  | 84.353 (39.021)
  Month 84: number analyzed (Participants) | 160 | 0 | 51
  Month 84 | 91.179 (38.381) |  | 87.673 (37.769)
  Month 90: number analyzed (Participants) | 103 | 0 | 44
  Month 90 | 84.206 (31.74) |  | 97.65 (38.203)
  Month 96: number analyzed (Participants) | 97 | 0 | 45
  Month 96 | 83.425 (34.159) |  | 98.767 (39.647)
  Month 108: number analyzed (Participants) | 76 | 0 | 0
  Month 108 | 79.499 (36.386) |  |
  Month 120: number analyzed (Participants) | 49 | 0 | 0
  Month 120 | 88.308 (41.251) |  |

10. Secondary Outcome: Changes in Endometrial Thickness Based on Transvaginal Ultrasonography at One Year, Five Years and Ten Years
Description: The Changes in Endometrial Thickness Based on Transvaginal Ultrasonography at One Year, Five Years and Ten Years.
Time Frame: 10 Years
Population: Endometrial thickness (ET) was evaluated in 52 LILETTA Efficacy Group subjects in the LNG20 (16-35 Yr Olds) arm only, with data both at Baseline and Month 12 (ET population) as part of a substudy conducted within the main protocol.
Measure: Mean (Standard Deviation); unit: Endometrial Thickness (mm)
Groups:
- LNG20: LNG20 levonorgestrel-releasing intrauterine system
  LNG20: levonorgestrel-releasing intrauterine system for contraception
Arm/Group | LNG20
Number analyzed (Participants) | 52
Endometrial Thickness (mm)
  Baseline | 4.0 (2.4)
  Month 12 | 3.8 (1.8)
  Month 60: number analyzed (Participants) | 22
  Month 60 | 3.1 (1.5)
  Month 120: number analyzed (Participants) | 5
  Month 120 | 2.6 (1.1)

11. Secondary Outcome: Ex Vivo Analysis of IUSs That Are Removed or Expelled During the Study
Description: Analysis of residual LNG content from an appropriate sampling of IUSs that were removed or expelled during the study was to be summarized and plotted as a function of time of removal/expulsion. Residual drug content analysis was performed on a sampling of removed or expelled samples to determine the average in vivo drug release rate during the time the samples were implanted. All available samples were sorted and grouped by duration of use in 90-day intervals. The drug content and time of exposure of the samples analyzed were fit by an exponential regression to calculate the initial and average in vivo release rate over the duration of the study.
  NOTE: Year = 360 day intervals
Time Frame: 8 Years
Population: In this substudy, a sampling of removed or expelled LNG20 IUSs were evaluated for residual drug content from Day 1 through Year 8. The total number of IUSs analyzed was 130 units from a total of 130 participants. All IUSs came from participants in the LNG20 (16-35 Yr Olds) arm. IUSs from participants in the Mirena arm were not evaluated in this substudy.
Measure: Mean (Standard Deviation); unit: mg/day
Units Other Than Participants: IUS
Arm/Group | LNG20
Number analyzed (Participants) | 130
Number analyzed (IUS) | 130
mg/day
  Year 1: number analyzed (Participants) | 28
  Year 1: number analyzed (IUS) | 28
  Year 1 | 45.1 (1.8)
  Year 2: number analyzed (Participants) | 24
  Year 2: number analyzed (IUS) | 24
  Year 2 | 39.1 (1.8)
  Year 3: number analyzed (Participants) | 18
  Year 3: number analyzed (IUS) | 18
  Year 3 | 33.8 (1.8)
  Year 4: number analyzed (Participants) | 12
  Year 4: number analyzed (IUS) | 12
  Year 4 | 29.3 (1.8)
  Year 5: number analyzed (Participants) | 12
  Year 5: number analyzed (IUS) | 12
  Year 5 | 25.4 (1.8)
  Year 6: number analyzed (Participants) | 12
  Year 6: number analyzed (IUS) | 12
  Year 6 | 22.0 (1.8)
  Year 7: number analyzed (Participants) | 12
  Year 7: number analyzed (IUS) | 12
  Year 7 | 19.1 (1.8)
  Year 8: number analyzed (Participants) | 12
  Year 8: number analyzed (IUS) | 12
  Year 8 | 16.6 (1.8)

12. Secondary Outcome: Incidence of Bleeding and/or Spotting
Description: From data based on the daily diary log, number of IUS subjects experiencing some bleeding and/or spotting.
Time Frame: 8 Years
Population: Any incidences of bleeding and/or spotting were self-reported via daily diary log by remaining participants at regular intervals throughout the length of the study. All Mirena participants were discontinued by the end of Year 5.
Measure: Count of Participants; unit: Participants
Arm/Group | LNG20 (16-35 Yr Olds) | Mirena | LNG20 (36-45 Yr Olds)
Number analyzed (Participants) | 1545 | 151 | 146
Participants
  Cycle 1 (Days 0- 28) | 1536 | 150 | 145
  Cycle 2 (Days 29 - 57): number analyzed (Participants) | 1509 | 145 | 146
  Cycle 2 (Days 29 - 57) | 1394 | 131 | 139
  Cycle 3 (Days 58 - 86): number analyzed (Participants) | 1486 | 143 | 143
  Cycle 3 (Days 58 - 86) | 1276 | 122 | 122
  Year 1: number analyzed (Participants) | 1320 | 123 | 128
  Year 1 | 1070 | 97 | 109
  Year 2: number analyzed (Participants) | 1062 | 81 | 114
  Year 2 | 779 | 54 | 79
  Year 3: number analyzed (Participants) | 876 | 65 | 105
  Year 3 | 557 | 44 | 65
  Year 4: number analyzed (Participants) | 743 | 51 | 97
  Year 4 | 468 | 28 | 60
  Year 5: number analyzed (Participants) | 618 | 38 | 89
  Year 5 | 369 | 22 | 54
  Year 6: number analyzed (Participants) | 509 | 0 | 78
  Year 6 | 310 |  | 45
  Year 7: number analyzed (Participants) | 417 | 0 | 72
  Year 7 | 260 |  | 39
  Year 8: number analyzed (Participants) | 304 | 0 | 61
  Year 8 | 189 |  | 33

13. Secondary Outcome: Cumulative Pregnancy Rates
Description: Life table methods were used to estimate the cumulative pregnancy rate after each year. Confirmed pregnancy was the failure outcome and the corresponding time to pregnancy was the failure time. Time to pregnancy was calculated as the date a confirmed pregnancy was initially reported minus the date of IUS placement plus one.
Time Frame: 8 years
Population: Note: a year is considered 364 days (13 women-months). Only the efficacy population (LNG20 16-35 years old) was evaluated, per protocol.
Measure: Number (95% Confidence Interval); unit: number of pregnancies per year
Groups:
- LNG20: No Cycles Excluded (MITT Population): LNG20 levonorgestrel-releasing intrauterine system LNG20: levonorgestrel-releasing intrauterine system for contraception with no cycles excluded
Arm/Group | LNG20: No Cycles Excluded (MITT Population)
Number analyzed (Participants) | 1545
number of pregnancies per year
  Year 1 | 0.14 [0.04 to 0.57]
  Year 2 | 0.49 [0.22 to 1.09]
  Year 3 | 0.59 [0.28 to 1.25]
  Year 4 | 0.72 [0.36 to 1.45]
  Year 5 | 0.87 [0.44 to 1.70]
  Year 6 | 0.87 [0.44 to 1.70]
  Year 7 | 1.30 [0.69 to 2.47]
  Year 8 | 1.30 [0.69 to 2.47]

14. Secondary Outcome: Expulsion Rate
Description: The expulsion rate includes the number of subjects with reported expulsions or removal of the IUS, regardless of reason.
Time Frame: 10 years
Population: All Mirena participants were discontinued by end of Year 5 per the study protocol. All LNG20 (36-45 Yr Old) participants were discontinued by end of Year 8 per the study protocol.
Measure: Count of Participants; unit: Participants
Arm/Group | LNG20 (16-35 Year Olds) | Mirena | LNG20 (36-45 Year Olds)
Number analyzed (Participants) | 1600 | 159 | 151
Participants
  IUS Placement through Year 1 | 47 | 8 | 3
  Year 1 through Year 2 | 5 | 4 | 1
  Year 2 through Year 3 | 2 | 0 | 0
  Year 3 through Year 4 | 2 | 1 | 2
  Year 4 through Year 5 | 1 | 0 | 0
  Year 5 through Year 6: number analyzed (Participants) | 1600 | 0 | 151
  Year 5 through Year 6 | 2 | 0 | 0
  Year 6 through Year 7: number analyzed (Participants) | 1600 | 0 | 151
  Year 6 through Year 7 | 2 | 0 | 1
  Year 7 through Year 8: number analyzed (Participants) | 1600 | 0 | 151
  Year 7 through Year 8 | 2 | 0 | 0
  Year 8 through Year 9: number analyzed (Participants) | 1600 | 0 | 0
  Year 8 through Year 9 | 1 | 0 | 0
  Year 9 through Year 10: number analyzed (Participants) | 1600 | 0 | 0
  Year 9 through Year 10 | 0 | 0 | 0

15. Secondary Outcome: Change in Hemoglobin Values
Description: Measuring the change in hemoglobin results from the screening visit and following 12 months, 60 months and 120 months of product use.
Time Frame: 10 years
Population: No standard deviation since there was only one Mirena participant measured at month 120
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | LNG20 (16-35 Yr Olds) | Mirena | LNG20 (36-45 Yr Olds)
Number analyzed (Participants) | 1600 | 159 | 151
g/dL
  Change from Screening to Month 12: number analyzed (Participants) | 1344 | 122 | 123
  Change from Screening to Month 12 | 0.2 (0.9) | 0.2 (1.1) | 0.1 (0.8)
  Change from Screening to Month 60: number analyzed (Participants) | 521 | 35 | 78
  Change from Screening to Month 60 | 0.3 (1.0) | 0.1 (1.1) | 0.3 (0.8)
  Change from Screening to Month 120: number analyzed (Participants) | 457 | 1 | 66
  Change from Screening to Month 120 | 0.3 (1.0) | -0.7 (NA) — No standard deviation since there was only one Mirena participant measured at month 120 | 0.3 (0.9)

16. Secondary Outcome: Discontinuation for Safety Reasons
Description: Time to event was calculated as the date of continuation/expulsion/removal minus the date of IUS placement plus one. Subjects without a continuation/expulsion/removal were censored at the last contact date and failure time was calculated as the last contact date minus the date of IUS placement plus one.
Time Frame: 10 years
Population: All Mirena participants were discontinued by end of Year 5 per the study protocol. All LNG20 (36-45 Yr Old) participants were discontinued by Year 8 per the study protocol.
Measure: Count of Participants; unit: Participants
Arm/Group | LNG20 (16-35 Yr Olds) | Mirena | LNG20 (36-45 Yr Olds)
Number analyzed (Participants) | 1600 | 159 | 151
Participants
  Year 1 | 5 | 3 | 0
  Year 2 | 0 | 0 | 0
  Year 3 | 1 | 0 | 0
  Year 4 | 0 | 0 | 0
  Year 5 | 0 | 0 | 0
  Year 6: number analyzed (Participants) | 1600 | 0 | 151
  Year 6 | 0 | 0 | 0
  Year 7: number analyzed (Participants) | 1600 | 0 | 151
  Year 7 | 0 | 0 | 0
  Year 8: number analyzed (Participants) | 1600 | 0 | 151
  Year 8 | 0 | 0 | 0
  Year 9: number analyzed (Participants) | 1600 | 0 | 0
  Year 9 | 0 | 0 | 0
  Year 10: number analyzed (Participants) | 1600 | 0 | 0
  Year 10 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: 10 years
Description: An Adverse Event (AE) was defined as any untoward medical occurrence in a patient or clinical investigation subject administered a pharmaceutical product and which does not necessarily have to have a causal relationship with this treatment. An AE could be any unfavorable and unintended sign (including a clinically significant abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product.
Arm/Group | LNG20 (16-35 Yr Olds) | Mirena | LNG20 (36-45 Yr Olds)
All-Cause Mortality (participants affected / at risk) | 1/1600 | 0/159 | 0/151
Serious Adverse Events (participants affected / at risk) | 78/1600 | 6/159 | 8/151
Other Adverse Events (participants affected / at risk) | 1441/1600 | 138/159 | 137/151
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | LNG20 (16-35 Yr Olds) (N=1600) | Mirena (N=159) | LNG20 (36-45 Yr Olds) (N=151)
Arnold-Chiari malformation (Congenital, familial and genetic disorders) | 1 | 0 | 0
Hamartoma (Congenital, familial and genetic disorders) | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 67 | 5 | 7
Colitis ulcerative (Gastrointestinal disorders) | 1 | 0 | 1
Crohn's disease (Gastrointestinal disorders) | 3 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 31 | 5 | 8
Enteritis (Gastrointestinal disorders) | 2 | 0 | 0
Oesophageal achalasia (Gastrointestinal disorders) | 0 | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 2 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 1 | 0
Catheter related complication (General disorders) | 1 | 0 | 0
Non-cardiac chest pain (General disorders) | 2 | 0 | 1
Bile duct obstruction (Hepatobiliary disorders) | 1 | 0 | 0
Cholecystitis (Hepatobiliary disorders) | 4 | 0 | 1
Cholecystitis acute (Hepatobiliary disorders) | 2 | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 7 | 4 | 2
Portal vein thrombosis (Hepatobiliary disorders) | 1 | 0 | 0
Anaphylactic reaction (Immune system disorders) | 3 | 0 | 0
Appendicitis (Infections and infestations) | 7 | 1 | 1
Appendix perforated (Infections and infestations) | 1 | 0 | 0
Cellulitis (Infections and infestations) | 14 | 0 | 3
Clostridial infection (Infections and infestations) | 5 | 2 | 0
Diverticulitis (Infections and infestations) | 2 | 1 | 0
Herpes Simplex (Infections and infestations) | 17 | 0 | 2
Lobar pneumonia (Infections and infestations) | 1 | 0 | 0
Pelvic inflammatory disease (Infections and infestations) | 9 | 0 | 0
Pneumonia streptococcal (Infections and infestations) | 1 | 0 | 0
Postoperative abscess (Infections and infestations) | 1 | 0 | 0
Respiratory tract infection (Infections and infestations) | 5 | 0 | 0
Tooth abscess (Infections and infestations) | 13 | 1 | 5
Ankle fracture (Injury, poisoning and procedural complications) | 3 | 0 | 0
Laceration (Injury, poisoning and procedural complications) | 2 | 0 | 0
Multiple drug overdose (Injury, poisoning and procedural complications) | 1 | 0 | 0
Pelvic fracture (Injury, poisoning and procedural complications) | 1 | 1 | 0
Rib fracture (Injury, poisoning and procedural complications) | 4 | 1 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 33 | 1 | 4
Traumatic liver injury (Injury, poisoning and procedural complications) | 1 | 0 | 0
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 46 | 5 | 8
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0
Chronic lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Dermatofibrosarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Ewing's sarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 0 | 1
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 2
Malignant melanoma stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Neoplasm of appendix (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Squamous cell carcinoma of the cervix (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Carotid artery thrombosis (Nervous system disorders) | 1 | 0 | 0
Intracranial hypotension (Nervous system disorders) | 1 | 0 | 0
Ischaemic stroke (Nervous system disorders) | 1 | 0 | 0
Multiple sclerosis (Nervous system disorders) | 6 | 0 | 0
Nervous system disorder (Nervous system disorders) | 1 | 0 | 0
Syncope (Nervous system disorders) | 22 | 0 | 1
Ectopic pregnancy (Pregnancy, puerperium and perinatal conditions) | 7 | 1 | 0
Affective disorder (Psychiatric disorders) | 2 | 0 | 0
Alcohol withdrawal syndrome (Psychiatric disorders) | 1 | 0 | 0
Bipolar I disorder (Psychiatric disorders) | 2 | 0 | 0
Bipolar disorder (Psychiatric disorders) | 15 | 4 | 1
Completed suicide (Psychiatric disorders) | 1 | 0 | 0
Delusional disorder, unspecified type (Psychiatric disorders) | 1 | 0 | 0
Drug abuse (Psychiatric disorders) | 2 | 0 | 0
Mania (Psychiatric disorders) | 1 | 0 | 1
Psychiatric symptom (Psychiatric disorders) | 1 | 0 | 0
Substance abuse (Psychiatric disorders) | 1 | 0 | 0
Suicidal ideation (Psychiatric disorders) | 4 | 0 | 0
Suicide attempt (Psychiatric disorders) | 2 | 0 | 0
Calculus ureteric (Renal and urinary disorders) | 2 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 14 | 1 | 6
Renal failure chronic (Psychiatric disorders) | 1 | 0 | 0
Renal vasculitis (Renal and urinary disorders) | 1 | 0 | 0
Ovarian cyst (Reproductive system and breast disorders) | 74 | 3 | 8
Ovarian cyst ruptured (Reproductive system and breast disorders) | 9 | 0 | 0
Ovarian torsion (Reproductive system and breast disorders) | 1 | 0 | 0
Vaginal laceration (Reproductive system and breast disorders) | 6 | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pulmonary Oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 0 | 1
Haematoma (Vascular disorders) | 0 | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Diaphragmatic hernia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Chronic respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Ovarian rupture (Reproductive system and breast disorders) | 0 | 1 | 0
Self-injurious ideation (Psychiatric disorders) | 0 | 1 | 0
Carotid artery dissection (Nervous system disorders) | 0 | 1 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 11 | 3 | 4
Traumatic lung injury (Injury, poisoning and procedural complications) | 0 | 1 | 0
Skull fractured base (Injury, poisoning and procedural complications) | 0 | 1 | 0
Extradural haematoma (Injury, poisoning and procedural complications) | 0 | 1 | 0
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 1 | 1 | 0
Gastritis (Gastrointestinal disorders) | 9 | 2 | 2
Anaemia (Blood and lymphatic system disorders) | 14 | 3 | 3
Coagulopathy (Blood and lymphatic system disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | LNG20 (16-35 Yr Olds) (N=1600) | Mirena (N=159) | LNG20 (36-45 Yr Olds) (N=151)
Nausea (Gastrointestinal disorders) | 127 | 11 | 8
Bronchitis (Infections and infestations) | 102 | 7 | 16
Influenza (Infections and infestations) | 168 | 17 | 13
Nasopharyngitis (Infections and infestations) | 386 | 27 | 22
Pharyngitis streptococcal (Infections and infestations) | 89 | 7 | 10
Sinusitis (Infections and infestations) | 179 | 17 | 16
Upper respiratory tract infection (Infections and infestations) | 191 | 18 | 24
Urinary tract infection (Infections and infestations) | 287 | 25 | 27
Vaginitis bacterial (Infections and infestations) | 283 | 23 | 32
Vulvovaginal mycotic infection (Infections and infestations) | 287 | 27 | 17
Human papilloma virus test positive (Investigations) | 88 | 5 | 9
Weight increased (Investigations) | 87 | 10 | 19
Back pain (Musculoskeletal and connective tissue disorders) | 98 | 6 | 15
Headache (Nervous system disorders) | 145 | 13 | 21
Anxiety (Psychiatric disorders) | 148 | 14 | 20
Depression (Psychiatric disorders) | 126 | 10 | 8
Breast tenderness (Reproductive system and breast disorders) | 123 | 10 | 10
Cervical dysplasia (Reproductive system and breast disorders) | 212 | 11 | 18
Dysmenorrhoea (Reproductive system and breast disorders) | 128 | 0 | 3
Dyspareunia (Reproductive system and breast disorders) | 125 | 4 | 3
Pelvic pain (Reproductive system and breast disorders) | 113 | 10 | 5
Vaginal discharge (Reproductive system and breast disorders) | 93 | 9 | 8
Acne (Skin and subcutaneous tissue disorders) | 247 | 20 | 12
Seasonal allergy (Immune system disorders) | 64 | 8 | 9
Insomnia (Psychiatric disorders) | 53 | 9 | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2017-10-02): https://cdn.clinicaltrials.gov/large-docs/50/NCT00995150/Prot_000.pdf
  • Statistical Analysis Plan (2017-10-02): https://cdn.clinicaltrials.gov/large-docs/50/NCT00995150/SAP_001.pdf